CLINICAL TRIAL: NCT06973720
Title: A Phase 2b, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy, Safety and Tolerability of Multiple Dose Regimens of Once-Weekly Switching to Once-Monthly MET097 in Participants With Obesity or Overweight (VESPER-3)
Brief Title: A Phase 2b Study to Evaluate the Efficacy and Safety of Once-Monthly MET097 in Adults With Obesity or Overweight
Acronym: VESPER-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Metsera, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET097-25-203
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight or Obesity
Keywords: Overweight; GLP-1
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MET097 (Experimental): Participants will be randomized to one of four dosing regimens receiving twelve weekly doses of MET097 (with or without titration) followed by multiple monthly doses.
  Interventions: Drug: MET097
- Placebo (Placebo Comparator): Participants who are randomized to the placebo arm will receive twelve weekly doses of placebo followed by multiple monthly doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MET097 — For subcutaneous administration.
  Arms: MET097
Drug: Placebo — Sterile 0.9% (w/v) saline for subcutaneous administration.
  Arms: Placebo

SUMMARY:
This study is designed to test the weight loss effects, safety, and tolerability of multiple monthly doses of MET097 after 12 weekly doses, compared to placebo. Participants are eligible if they have overweight or obesity and do not have type 2 diabetes.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study to investigate the efficacy, safety and tolerability of multiple once monthly (QM) dose levels of MET097 after 12 once weekly (QW) doses, compared to placebo. The study will include adult participants with obesity or overweight. Participants will initially receive once weekly MET097 with or without titration or placebo for 12 weeks. Participants will then transition to a four-fold higher monthly dose for a total of 13 monthly doses. The primary endpoint is at Week 28, four weeks after the fourth monthly dose. All participants will be followed for ~5 half-lives after administration of the last dose for safety.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) at Screening of:

  * BMI ≥30 kg/m2 and ≤50.0 kg/m2 (can have the weight-related co-morbidities listed below)
  * BMI ≥27.0 kg/m2 to <30.0 kg/m2 with at least one of the following weight-related co-morbidities:

    1. Hypertension: on blood pressure (BP)-lowering medication or having systolic BP ≥130 mmHg or diastolic BP ≥80 mmHg at Screening
    2. Dyslipidemia: on lipid-lowering medication or having low-density lipoprotein cholesterol (LDL-C) ≥160 mg/dL (4.1 mmol/L) or triglycerides ≥150 mg/dL (1.7 mmol/L), or high-density lipoprotein-cholesterol (HDL-C) <40 mg/dL (1.0 mmol/L) for men or HDL-C <50 mg/dL (1.3 mmol/L) for women at Screening
    3. Stable body weight (increase or decrease ≤5 kg) within 3 months prior to Screening

Exclusion Criteria:

* Diagnosis of diabetes (T1DM or T2DM) or glycated hemoglobin A1c (HbA1c) ≥ 6.5% or fasting plasma glucose >125 mg/dL.
* Estimated glomerular filtration rate (eGFR) <75 mL/min/1.73 m2
* History of pancreatitis
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Poorly controlled hypertension at, defined as any of the following:

  * Mean seated systolic BP ≥160 mm Hg or mean seated diastolic BP ≥95 mm Hg at Screening visit
  * A change in antihypertensive medications within 30 days of Screening visit
  * Renal artery stenosis, or evidence of labile blood pressure including symptomatic postural hypotension at Screening; postural hypotension is defined as a sustained reduction of systolic blood pressure of at least 20 mmHg or diastolic blood pressure of 10 mmHg, with or without symptoms during the assessment, within three minutes of standing
* Thyroid-stimulating hormone (TSH) level lower than 0.4 mIU/L or higher than 6.0 mIU/L at the Screening visit. Note: participants receiving treatment for hypothyroidism may be included, provided their thyroid hormone replacement dose has been stable for at least 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight at Week 28 | Baseline (Week 0) through Week 28 (Day 197)
  Evaluate the efficacy at Week 28 of four dose regimens of QW MET097 switching to QM compared to placebo.

SECONDARY OUTCOMES:
Percent change from baseline in body weight at Week 64 | Baseline (Week 0) through Week 64 (Day 449)
Percent change from baseline in body weight at all other post-baseline weight measurements up to Week 64 other than Week 28 | Baseline (Week 0) through Week 24 (Day 169); Week 32 (Day 225) through Week 64 (Day 449)
Change from baseline in absolute bodyweight (in kg) at all protocol-specified weekly and monthly post-baseline measurements | Baseline (Week 0) through Week 64 (Day 449)
Change from baseline in body mass index (BMI) at all protocol-specified weekly and monthly post-baseline measurements | Baseline (Week 0) through Week 64 (Day 449)
Change from baseline in waist circumference (in cm) at all protocol-specified weekly and monthly post-baseline measurements | Baseline (Week 0) through Week 64 (Day 449)
Percent change from baseline in body weight at post-treatment follow-up | Baseline (Week 0) through Week 72 (Day 505)
Change from baseline in absolute bodyweight (in kg) at post-treatment follow-up | Baseline (Week 0) through Week 72 (Day 505)
Change from baseline in body mass index (BMI) at post-treatment follow-up | Baseline (Week 0) through Week 72 (Day 505)
Change from baseline in waist circumference (in cm) at post-treatment follow-up | Baseline (Week 0) through Week 72 (Day 505)
Occurrence of treatment emergent adverse events (TEAEs) | Baseline (Week 0) through Week 72 (Day 505)
Minimum observed concentration (Cmin) | Baseline (Week 0) through Week 72 (Day 505)
Area under the concentration versus time curve during the dosing interval (AUC) | Baseline (Week 0) through Week 72 (Day 505)
Maximum observed concentration (Cmax) | Baseline (Week 0) through Week 72 (Day 505)
Time to maximum concentration (Tmax) | Baseline (Week 0) through Week 72 (Day 505)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Research Site 097203-001001, Hollywood, Florida
  - Research Site 097203-001003, Tampa, Florida
  - Research Site 097203-001002, Decatur, Georgia
  - Research Site 097203-001005, Savannah, Georgia
  - Research Site 097203-001004, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided